CLINICAL TRIAL: NCT06097832
Title: Phase 1b/2 Study of NXC-201 for the Treatment of Patients With Relapsed or Refractory AL Amyloidosis
Brief Title: Study of NXC-201 CAR-T in Patients With Light Chain (AL) Amyloidosis
Acronym: NEXICART-2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nexcella Inc. (Industry)
Collaborators: Immix Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NXC-201-AL-001
Record Dates: First submitted 2023-10-14; First posted 2023-10-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-01

CONDITIONS: Light Chain (AL) Amyloidosis
Keywords: Relapsed refractory AL amyloidosis; R/R AL amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Intervention Model Description: Open label single-arm clinical study of NXC-201 CAR-T will proceed sequentially through dose cohorts as follows:
  Cohort 1 - 150×10^6 CAR-positive (CAR+) T cells (3 patients)
  Cohort 2 - 450×10^6 CAR-positive (CAR+) T cells (3 patients)
  The dose expansion phase will then proceed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NXC-201 CAR-T (Experimental): The dose escalation phase will include the following doses:
  Cohort 1 - 150×10^6 CAR-positive (CAR+) T cells (3 patients) Cohort 2 - 450×10^6 CAR-positive (CAR+) T cells (3 patients) The dose expansion phase will then proceed.
  Interventions: Biological: NXC-201 CAR-T

INTERVENTIONS:
Biological: NXC-201 CAR-T — NXC-201 (formerly HBI0101) CAR-T is defined as autologous T cells transduced ex-vivo with anti-BCMA CAR retroviral vector encoding the chimeric antigen receptor (CAR) targeted to human BCMA. The NXC-201 CAR-T is provided fresh without cryopreservation.
  Other Names: HBI0101 CAR-T

SUMMARY:
Open-label Phase 1b Dose Escalation/Dose Expansion study exploring the safety and efficacy of NXC-201 in patients with relapsed or refractory light chain amyloidosis (AL).

DETAILED DESCRIPTION:
Building on the prior NXC-201 results in AL amyloidosis published by Kfir-Erenfeld et. al (2022) and Asherie et. al. (2023), this study will enroll additional patients with relapsed or refractory AL amyloidosis and assess the safety and efficacy of NXC-201.

Subjects with relapsed/refractory AL amyloidosis will undergo leukapheresis at least one month prior to lymphodepletion, to provide starting material for NXC-201 CART manufacture. Subjects will be treated according to the following process for lymphodepletion: Days -5, -4 and -3 Cyclophosphamide 250mg/m2, IV infusion over 30 mins, followed immediately by Fludarabine 25 mg/m2 IV infusion over 30 minutes.

NXC-201 CART is administered on Day 0, after lymphodepletion.

Enrolled subjects will receive a dose of NXC-201 CAR-positive (CAR+) T cells. Dose escalation and expansion will be guided by safety review committee.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Voluntarily signed informed consent form (ICF).
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
4. Histologically proven systemic AL amyloidosis confirmed by positive Congo red staining with green birefringence on polarized light microscopy in an organ outside the bone marrow and evidence of a measurable clonal plasma cell disease that requires active treatment.

   1. An underlying plasma cell disorder can be identified by one of the following: clonal plasma cells in the BM, monoclonal protein in the serum or urine, or abnormal free light chain ratio.
   2. Because AL amyloidosis may present with low volumes of bone marrow plasma cells, prior biopsies demonstrating clonal plasma cell populations may be used to determine eligibility.
   3. Measurable hematologic disease: difference between involved and uninvolved FLC > 20 mg/L (or 2mg/dl) with an abnormal k/l ratio; or M-spike > 0.5mg/dl.
5. Patients should have received at least one line of therapy with a CD38 monoclonal antibody and a proteosome inhibitor and not be in VGPR or CR at the time of inclusion. Patients who did not reach VGPR after two cycles of initial therapy or patients who did achieve VGPR or better but with a hematological relapse can be included.
6. Symptomatic organ involvement (heart, kidney, liver/GI tract, peripheral nervous system).
7. Women of child-bearing potential (WCBP) must have a negative serum pregnancy test prior to treatment. All sexually active WCBP and all sexually active male subjects must agree to use effective methods of birth control throughout the study.
8. Recovery to ≤Grade 2 or baseline of any non-hematologic toxicities due to prior treatments, excluding alopecia and Grade 3 neuropathy.
9. Absence of any psychological, familial, sociological, or geographical conditions potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before trial entry.
10. Able to swallow pills.

Exclusion Criteria:

1. Prior treatment with CAR T therapy directed at any target.
2. Any therapy that is targeted to BCMA.
3. Stroke or seizure within 6 months of signing ICF.
4. Bone marrow plasma cells >30% and clinically symptomatic multiple myeloma with end organ damage (i.e. lytic bone lesions).
5. New York Heart Association Heart Failure Class III or Class IV.
6. Any prior systemic therapy for AL amyloidosis within 14 days prior to leukapheresis.
7. Therapeutic doses of steroids within 2 weeks prior to leukapheresis (Physiological replacement doses of steroids are allowed up to 12 mg/m2/d hydrocortisone or equivalent).
8. Any prior systemic therapy for AL amyloidosis within 14 days of leukapheresis.
9. Wash-out period of at least 4 weeks from previous investigational treatment prior to leukapheresis.
10. Inadequate hepatic function:

    1. Aspartate aminotransferase (AST [SGOT] or alanine aminotransferase (ALT [SGPT]) >3 x upper limit of normal (ULN) value
    2. Alkaline phosphatase >2 times ULN
    3. Serum direct bilirubin >2 times ULN
11. Inadequate renal function: creatinine clearance (CRCL) <20 mL/min.
12. International ratio (INR) or partial thromboplastin time (PTT) >1.5 x ULN, unless on a stable dose of anticoagulant for a thromboembolic event that does NOT meet exclusion criteria.
13. Inadequate bone marrow function prior to leukapheresis or lymphodepletion, without transfusion or growth factor support within 5 days prior defined by absolute neutrophil count (ANC) <1000 cells/mm3, platelet count <50,000/mm3, or hemoglobin <8 g/dL (blood transfusions are allowed), absolute lymphocyte count < 300 cells/mm3.
14. Presence of active infection within 72 hours prior to lymphodepletion.
15. Significant co-morbid condition/s or disease/s which in the judgment of the Investigator would place the subject at undue risk or interfere with the study.
16. Known human immunodeficiency virus (HIV) positive status subjects who have not achieved undetectable viral load on highly active anti-retroviral therapy/combination anti-retroviral therapy (HAART/cART) within 6 months of lymphodepletion (previously treated HIV with undetectable viral load can be included)
17. Patients with active Hepatitis B or Hepatitis C with detectable viral load (previously treated Hepatitis B or Hepatitis C with undetectable viral load can be included)
18. Subjects with a history of stroke, unstable angina, or myocardial infarction requiring medication or mechanical control within 3 months.
19. Evidence of clinically significant ventricular arrhythmias on 7-day Zio® patch (or equivalent device) monitoring despite anti-arrhythmic treatment, except if a pacemaker or automated implantable cardioverter defibrillator (AICD) has been implanted.
20. Stage IIIb patients:

    1. NT-proBNP >8500 ng/L and
    2. hs-troponin I ≥100 ng/L or troponin I ≥0.1 mcg/L or troponin T ≥ 0.035 mcg/L or hs-troponin T ≥50 ng/L
21. Left ventricular ejection fraction <35%.
22. Heart failure which is, in the opinion of the Investigator, related to ischemic heart disease.
23. Presence of other active malignancy that requires treatment with the exception of non-melanoma skin cancer, cervical cancer, treated early-stage prostate cancer provided that prostate specific antigen is within normal limit, or any completely resected carcinoma in situ; other indolent/completely resected malignancies may be discussed with the Principal Investigator (PI) and/or Co-PI.
24. Subjects who have had a venous thromboembolic event requiring anticoagulation and who meet any of the following criteria:

    1. Have been on a stable dose of anticoagulation for < 1 month (except for acute line insertion induced thrombosis).
    2. Have had a Grade 2, 3, or 4 hemorrhage in the last 30 days.
    3. Are experiencing continued symptoms from their venous thromboembolic event (e.g., continued dyspnea or oxygen requirement).
25. Presence of non-AL amyloidosis.
26. AL amyloidosis with isolated soft tissue involvement.
27. Supine systolic blood pressure <100 mmHg or postural symptoms despite medical therapy.
28. Subject is a woman who is pregnant, or breast-feeding, or planning to become pregnant.
29. Subjects with known/underlying medical conditions that, in the investigator's opinion would make the administration of the study drug hazardous (i.e., chronic obstructive pulmonary disease, persistent asthma, uncontrolled diabetes or uncontrolled coronary artery disease).
30. Chronic atrial fibrillation with uncontrolled heart rate.
31. Unwillingness to practice effective birth control.
32. Inability to comply with other requirements of the protocol.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2039-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | 24 months
  An adverse event (AE) can be any unfavorable and unintended sign (including an abnormal. laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Number of Participants with Adverse Events by Severity as Assessed by CTCAE v5.0 | 24 months
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0, with the exception of cytokine release syndrome (CRS), and immune effector cell-associated neurotoxicity syndrome (ICANS). CRS and ICANS should be evaluated according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading.
To confirm the maximum tolerated dose (MTD) | 24 months
  According to Common Terminology Criteria for Adverse Events (CTCAE) criteria, version 5.0, and Cytokine release syndrome (CRS) and Immune effector cell-associated neurotoxicity syndrome (ICANS) per American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading
To confirm the recommended phase 2 dose (RP2D) | 24 months
  According to Common Terminology Criteria for Adverse Events (CTCAE) criteria, version 5.0, and Cytokine release syndrome (CRS) and Immune effector cell-associated neurotoxicity syndrome (ICANS) per American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading

SECONDARY OUTCOMES:
Percentage of participants with hematologic and organ response | 24 months
  According to consensus recommendations for AL amyloidosis treatment response criteria in AL (Palladini, 2012)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Sutter Health Alta Bates, Berkeley, California
  - City of Hope, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Stanford University, Stanford, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - The University of Kansas Cancer Center, Fairway, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Comprehensive Cancer Center, New York, New York
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
There will be no individual participant data sharing

REFERENCES:
- [Background] Kfir-Erenfeld S, Asherie N, Grisariu S, Avni B, Zimran E, Assayag M, Sharon TD, Pick M, Lebel E, Shaulov A, Cohen YC, Avivi I, Cohen CJ, Stepensky P, Gatt ME. Feasibility of a Novel Academic BCMA-CART (HBI0101) for the Treatment of Relapsed and Refractory AL Amyloidosis. Clin Cancer Res. 2022 Dec 1;28(23):5156-5166. doi: 10.1158/1078-0432.CCR-22-0637. PMID 36107221
- [Background] Asherie N, Kfir-Erenfeld S, Avni B, Assayag M, Dubnikov T, Zalcman N, Lebel E, Zimran E, Shaulov A, Pick M, Cohen Y, Avivi I, Cohen C, Gatt ME, Grisariu S, Stepensky P. Development and manufacture of novel locally produced anti-BCMA CAR T cells for the treatment of relapsed/refractory multiple myeloma: results from a phase I clinical trial. Haematologica. 2023 Jul 1;108(7):1827-1839. doi: 10.3324/haematol.2022.281628. PMID 36200421
- [Background] Palladini G, Dispenzieri A, Gertz MA, Kumar S, Wechalekar A, Hawkins PN, Schonland S, Hegenbart U, Comenzo R, Kastritis E, Dimopoulos MA, Jaccard A, Klersy C, Merlini G. New criteria for response to treatment in immunoglobulin light chain amyloidosis based on free light chain measurement and cardiac biomarkers: impact on survival outcomes. J Clin Oncol. 2012 Dec 20;30(36):4541-9. doi: 10.1200/JCO.2011.37.7614. Epub 2012 Oct 22. PMID 23091105